CLINICAL TRIAL: NCT00423332
Title: A Phase II, Randomised, Double-blind, Parallel Group Study to Assess the Efficacy of Cediranib 45mg Versus Placebo Following 12 Weeks of Treatment in Patients With Metastatic or Recurrent Renal Cell Carcinoma Who Have Had no Previous Anti-VEGF Therapy.
Brief Title: Cediranib (AZD2171, RECENTIN™) in Metastatic or Recurrent Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00030; EudraCT no. 2006-002455-33
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-11

CONDITIONS: Renal Cell Carcinoma
Keywords: cancer; tumour; advanced cancer; Metastatic renal cell carcinoma; kidney cancer; RECENTIN
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Kidney Neoplasms | interventions — cediranib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator): Cediranib placebo
  Interventions: Drug: Cediranib Placebo
- 2 (Experimental): Cediranib
  Interventions: Drug: Cediranib

INTERVENTIONS:
Drug: Cediranib — 45 mg oral tablet
  Other Names: AZD2171; RECENTIN™
  Arms: 2
Drug: Cediranib Placebo — oral tablet
  Arms: 1

SUMMARY:
Cediranib is being tested to assess its effectiveness on the growth of kidney cancer tumours and also how well it is tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of metastatic or recurrent renal cell carcinoma

Exclusion Criteria:

* Certain types of previous anti-cancer therapy for Renal Cell Carcinoma
* Patients with type I insulin-dependent diabetes or poorly-controlled type II insulin-independent diabetes
* Patients with a history of poorly controlled high blood pressure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca
Locations (8):
- Netherlands (3):
  - Research Site, Groningen
  - Research Site, Leiden
  - Research Site, Nijmegen
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Oxford

REFERENCES:
- [Derived] Mulders P, Hawkins R, Nathan P, de Jong I, Osanto S, Porfiri E, Protheroe A, van Herpen CM, Mookerjee B, Pike L, Jurgensmeier JM, Gore ME. Cediranib monotherapy in patients with advanced renal cell carcinoma: results of a randomised phase II study. Eur J Cancer. 2012 Mar;48(4):527-37. doi: 10.1016/j.ejca.2011.12.022. Epub 2012 Jan 28. PMID 22285180
- See also: CSR-D8480C00030.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=419&filename=CSR-D8480C00030.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-one patients were randomised to study treatment: 53 to cediranib 45 mg and 18 to placebo. Following unblinding for the primary analysis, all patients, except those who had progressed on cediranib, then had the option of receiving open-label treatment with cediranib. Randomised=ITT=Safety set: Cediranib 45mg 53, Placebo 18.
Groups:
- AZD2171 45 mg: AZD2171 45mg/Day: 53 patients randomised
- Placebo: Placebo / Day: 18 patients randomised
Period: Overall Study
Arm/Group | AZD2171 45 mg | Placebo
Started | 53 (Randomised) | 18 (Number randomised)
Continuing After Unblinding | 44 (Number starting/ continuing AZD2171 after unblinding) | 14 (Number starting/ continuing AZD2171 after unblinding)
Ongoing at Data Cut Off (8th March 2009) | 22 (Number ongoing at data cut off (8th March 2009)) | 4 (Number ongoing at data cut off (8th March 2009))
Completed | 44 (Number completing 12 weeks blinded randomised treatment) | 11 (Number completing 12 weeks blinded randomised treatment)
Not Completed | 9 | 7
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Condition under investigation worsened | 1 | 1
Not completed — Progressive at Week 6 | 0 | 1
Not completed — Unblinded before 12 weeks | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- AZD2171 45 mg: AZD2171 45mg/Day
- Placebo: Placebo/Day
- Total: Total of all reporting groups
Arm/Group | AZD2171 45 mg | Placebo | Total
Number analyzed (Participants) | 53 | 18 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at informed consent
  Years | 60.7 (7.7) | 62.4 (8.7) | 61.2 (7.9)
Gender [Count of Participants; unit: Participants] — Gender at informed consent
  Participants
    Female | 13 | 3 | 16
    Male | 40 | 15 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Tumour Size at 12 Weeks
Description: Sum of longest diameters of the target lesions, based on Response Evaluation Criteria in Solid Tumours (RECIST) criteria ((Week 12 - baseline)/baseline)*100
Time Frame: Baseline to Week 12
Population: For patients to be included in the analysis they had to have been evaluable for RECIST with week 12 or progression tumour size data
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | AZD2171 45 mg | Placebo
Number analyzed (Participants) | 51 | 17
Percentage change from baseline | -19.47 (17.093) | 19.65 (22.902)

2. Secondary Outcome: Best Percentage Change From Baseline in Tumour Size During the Study
Description: Maximum reduction or minimum increase in tumour size where size is the sum of the longest diameters of the target lesions
Time Frame: Treatment period up to Week 12 visit date for last patient in (LPI)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | AZD2171 45 mg | Placebo
Number analyzed (Participants) | 51 | 17
Percentage change from baseline | -26.90 (23.153) | 1.09 (26.783)

3. Secondary Outcome: Duration of Response
Description: Based on RECIST measurements taken throughout the study and best objective tumour response at the defined analysis cut-off point. Measured from the time the criteria for complete response (CR)/partial response (PR) are first met (whichever is recorded first) until the patient progresses or dies.
Time Frame: Treatment period up to 2nd data cut-off of 8th March 2009
Population: For patients to be included in the analysis they had to have been evaluable for RECIST and have been a responder (Complete response (CR) or Partial Response (PR)).
  13 of the 19 responders had not progressed by the data cut off so their responses are ongoing and are censored at the date of the last evaluable visit before the data cut-off.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | AZD2171 45 mg | Placebo
Number analyzed (Participants) | 18 | 1
Months | 18.595 [12.517 to 18.595] | 11.1 [11.1 to 11.1]

4. Secondary Outcome: Progression Free Survival
Description: Number of months from randomisation until progressive disease based on RECIST (progression of target lesions, clear progression of existing non-target lesions or the appearance of one or more new lesions) or death in the absence of progression.
Time Frame: Treatment period up to 2nd data cut-off of 8th March 2009.
Population: Comparison of PFS between patients randomised to cediranib 45 mg versus those randomised to placebo. All patients irrespective of whether they had a 12 week scan are included in this analysis. At week 12 placebo patients were able to switch to cediranib.
Measure: Median (Full Range); unit: Months
Arm/Group | AZD2171 45 mg | Placebo
Number analyzed (Participants) | 53 | 18
Months | 12.1 [0 to 21.6] | 2.76 [0 to 21.5]

5. Secondary Outcome: Objective Tumour Response at 12 Weeks
Description: Number of patients with complete (CR) /partial response (PR) (based on RECIST). CR is defined as Disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of Longest Diameter (LD) of target lesions taking as reference the baseline sum LD. At 12 weeks, tumour responses would be unconfirmed, as this was the first post-baseline RECIST assessment, unless a patient had a RECIST assessment before Week 12 to confirm a suspected progression.
Time Frame: Response rate at 12 weeks was based on RECIST measurements taken at baseline and at Week 12, or upon progression if this was before Week 12.
Measure: Number; unit: Participants
Arm/Group | AZD2171 45 mg | Placebo
Number analyzed (Participants) | 53 | 18
Participants | 11 | 0

6. Secondary Outcome: Best Objective Tumour Response
Description: Best Objective Tumour response as defined by RECIST. Patients were assigned to 1 of the following best objective tumour response categories: complete response (CR) defined as a Disappearance of all target lesions, partial response (PR), defined as At least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD, stable disease (SD) defined as Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started, or progressive disease (PD) defined as At least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded (either at baseline or at previous assessment since treatment began). Patients who were evaluable for RECIST assessments, but who did not meet the criteria for CR, PR, SD, or PD, were assigned to the response category of not evaluable (NE).
Time Frame: Baseline, Week 12 and every 8 weeks thereafter or until progression.
Population: For the patients who switched from placebo to cediranib after unblinding, the baseline RECIST assessment was not reset to their last scan placebo, owing to the methods of data collection; therefore, it was not possible to determine their subsequent response to cediranib treatment using a 'best response' summary.
Measure: Number; unit: Participants
Arm/Group | AZD2171 45 mg | Placebo
Number analyzed (Participants) | 53 | 18
Participants | 18 | 1

ADVERSE EVENTS:
Groups:
- Cediranib DB; Placebo DB: Double Blind part
- Cediranib OL: Open Label part
Arm/Group | Cediranib DB | Placebo DB | Cediranib OL
Serious Adverse Events (participants affected / at risk) | 10/53 | 3/18 | 15/58
Other Adverse Events (participants affected / at risk) | 53/53 | 16/18 | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib DB (N=53) | Placebo DB (N=18) | Cediranib OL (N=58)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Calcium Increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1
Coma (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Loss Of Consciousness (Nervous system disorders) | 1 | 0 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1
Bartholin's Cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib DB (N=53) | Placebo DB (N=18) | Cediranib OL (N=58)
Splinter Haemorrhages (Cardiac disorders) | 3 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 0 | 2
Hypothyroidism (Endocrine disorders) | 4 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 39 | 5 | 35
Nausea (Gastrointestinal disorders) | 17 | 5 | 26
Constipation (Gastrointestinal disorders) | 16 | 4 | 10
Stomatitis (Gastrointestinal disorders) | 16 | 2 | 13
Vomiting (Gastrointestinal disorders) | 9 | 4 | 13
Abdominal Pain (Gastrointestinal disorders) | 7 | 2 | 9
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 0 | 3
Dry Mouth (Gastrointestinal disorders) | 3 | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 3
Glossodynia (Gastrointestinal disorders) | 3 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 3
Oral Pain (Gastrointestinal disorders) | 3 | 0 | 3
Toothache (Gastrointestinal disorders) | 3 | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 31 | 9 | 25
Feeling Cold (General disorders) | 5 | 0 | 0
Oedema Peripheral (General disorders) | 5 | 2 | 4
Chills (General disorders) | 3 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 1 | 2
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 5
Lower Respiratory Tract Infection (Infections and infestations) | 4 | 2 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 3
Oral Candidiasis (Infections and infestations) | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 1 | 1
Oral Herpes (Infections and infestations) | 0 | 1 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Weight Decreased (Investigations) | 6 | 1 | 15
Anorexia (Metabolism and nutrition disorders) | 13 | 0 | 11
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 0 | 11
Appetite Disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 8
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 24 | 4 | 10
Dizziness (Nervous system disorders) | 8 | 0 | 6
Lethargy (Nervous system disorders) | 7 | 1 | 2
Dysgeusia (Nervous system disorders) | 5 | 0 | 4
Paraesthesia (Nervous system disorders) | 1 | 1 | 4
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 0 | 4
Depression (Psychiatric disorders) | 1 | 0 | 5
Anxiety (Psychiatric disorders) | 2 | 1 | 0
Confusional State (Psychiatric disorders) | 2 | 1 | 2
Proteinuria (Renal and urinary disorders) | 4 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 31 | 1 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 11 | 0 | 12
Rash (Skin and subcutaneous tissue disorders) | 10 | 2 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash Erythematous (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 34 | 4 | 7
Flushing (Vascular disorders) | 3 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.